CLINICAL TRIAL: NCT06255145
Title: Assessment of Body Composition, Fatigue, Mobility and Functional Status in Post-Stroke Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Raziye ÇELİK, Principal Investigator physiotherapist, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: PamukkaleUniversityRC
Record Dates: First submitted 2023-10-14; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Cerebrovascular Stroke; Body Composition
Keywords: Stroke; Body Composition; Fatique; Mobility; Functional Status
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Based on the results of the power analysis, it was calculated that 80% power could be obtained at 95% confidence level when at least 42 people (21 people for each group) were included in the study all participants, body composition evaluation was carried out with the Beurer BF 1000 Super Precision device using the Bioelectrical Impedance Analysis principle, fatigue evaluation was carried out with the Fatigue Severity Scale, mobility evaluation was carried out with the Rivermead Mobility Index, and functional status evaluation was carried out with the Functional Independence Scale.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In all participants, body composition evaluation was carried out with the Beurer BF 1000 Super Precision device using the Bioelectrical Impedance Analysis principle, fatigue evaluation was carried out with the Fatigue Severity Scale, mobility evaluation was carried out with the Rivermead Mobility Index, and functional status evaluation was carried out with the Functional Independence Scale.
  Interventions: Device: Bioelectrical Impedance Analysis
- Control Group (Active Comparator): In all participants, body composition evaluation was carried out with the Beurer BF 1000 Super Precision device using the Bioelectrical Impedance Analysis principle, fatigue evaluation was carried out with the Fatigue Severity Scale, mobility evaluation was carried out with the Rivermead Mobility Index, and functional status evaluation was carried out with the Functional Independence Scale.
  Interventions: Device: Bioelectrical Impedance Analysis

INTERVENTIONS:
Device: Bioelectrical Impedance Analysis — Bioelectrical Impedance Analysis Beurer BF 1000 Super Precision device was used to measure the body composition of the participants. Operating on the principle of BIA, the device allows the body composition to be evaluated by giving an imperceptible electric current to the body.
  Fatigue Severity Scale (FSS) Fatigue Severity Scale (FSS) was used to measure participants' fatigue levels. Rivermead Mobility Index Rivermead Mobility Index (RMI) was used to assess the mobility levels of the participants.
  Functional Independence Measure Functional Independence Measure (FIM) was used to evaluate the functional status of the participants.
  Other Names: Fatigue Severity Scale; Rivermead Mobility Index; Functional Independence Scale

SUMMARY:
The goal of this randomized controlled trial is to evaluate body composition, fatigue, mobility level, functional status in with stroke individuals. The main questions it aims to answer are:

How is body composition affected in individuals with stroke? How is the level of fatigue affected in individuals with stroke? How is the mobility level affected in individuals with stroke? How is functional status affected in individuals with stroke? In this study, we included 21 patients with stroke and 21 healthy controls. The body composition of the participants was evaluated by Bioelectrical Impedance Analysis (BIA), fatigue level by Fatigue Severity Scale (FSS), mobility level by Rivermead Mobility Index (RMI), and functional status by Functional Independence Scale (FIM).

DETAILED DESCRIPTION:
As defined by the World Health Organization, stroke is "a clinical condition that has no apparent cause other than vascular causes, lasts for 24 hours or longer, or may result in death, and is characterized by sudden focal (or global) disturbances in cerebral function. It is the third leading cause of mortality in the world after cardiovascular diseases and cancer, and ranks first in terms of causing disability.¹ In Turkey, the incidence of stroke was estimated as 125,345 (154 per hundred thousand), the prevalence as 1,080,380 (1.3 percent), the mortality rate due to stroke as 48,947 people and the number of years of life lost due to stroke-related death/disability as 993,082 years.2Approximately 795000 people have a stroke in the United States of America every year and 185000 of them relapse.3 In 2016, stroke was responsible for approximately 5.5 million deaths and 116.4 million years of quality of life loss, with a significant impact on the economy.4 Post-stroke dysphagia, visual-spatial disorientation, gastrointestinal system disorders, depression, and increased catabolic process lead to malnutrition.5 In addition to hormonal changes and immobilization, fat mass increases while lean body mass decreases in individuals with stroke (IVS).6 Besides, following stroke, factors such as inadequate calorie and macronutrient intake, denervation, disuse, spasticity, and inflammation may come together to cause sarcopenia and thereby an increase in fat mass.5,7 Additionally, the study by Li et al. concluded that muscle loss after stroke is also accompanied by an increase in intramuscular fat and bone loss.8 In IVS, loss of muscle mass causes fatigue, general weakness and lack of energy. In one study, it was stated that skeletal muscle mass should be increased to reduce fatigue in IVS.9 Fatigue is a subjectively reported lack of physical and mental energy that negatively affects daily life activities. Among stroke survivors, 40% identified fatigue as one of the worst symptoms.10 IVS have gait and balance disorders due to motor, visual-perceptual, sensory problems, spasticity, paralysis, muscle atrophy, increase in fat mass, fatigue, movement limitations, proprioceptive sensory loss and impairments in cognitive functions. This situation can negatively affect the functional status of individuals by reducing their mobility levels.11,12 In stroke rehabilitation, it is important to identify the fat mass in individuals with stroke, to determine the loss of muscle mass in parallel, to determine in which regions the fat mass level increases more significantly, and to compare the fatigue and functional losses that may occur with this increase with healthy individuals in the same age group. In the literature, we did not find any study that evaluated body composition changes, fatigue, mobility and functional status together in IVS. The present study is significant in terms of examining the body composition of IVS in detail and evaluating the extent to which body composition parameters, fatigue, mobility and functional independence levels differ when compared with healthy controls. The purpose of our study is to compare body composition, fatigue, mobility and functional status in stroke patients with healthy subjects.

ELIGIBILITY:
Inclusion criteria for individuals with stroke:

* Being between the ages of 18-65
* Volunteering to participate in the study
* Having a score of 25 or above on the Mini Mental Test
* Getting a score between 0-3 on the Modified Rankin Scale

Exclusion criteria for individuals with stroke:

* Having cardiac insufficiency
* Being morbid obesity
* Having pacemaker
* Being pregnant

Inclusion criteria for healty individuals:

* Being between the ages of 30-65
* Volunteering to participate in the study
* Not having any neurological, orthopedic, rheumatologic and metabolic problems
* Having a score of 25 or above on the Mini Mental Test

Exclusion criteria for healty individuals:

* Participating in any fat burning diet program
* Exercising regularly
* Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Bioelectrical Impedance Analysis | 12 week
  body weight
Bioelectrical Impedance Analysis | 12 week
  body fat percentage
Bioelectrical Impedance Analysis | 12 week
  muscle percentage
Bioelectrical Impedance Analysis | 12 week
  total water percentage
Bioelectrical Impedance Analysis | 12 week
  visceral fat amount
Bioelectrical Impedance Analysis | 12 week
  total bone mass

SECONDARY OUTCOMES:
Fatigue Severity Scale | 12 week
  fatique. Minimum score is 9 and maximum score is 63. Scores of 36 or more represent severe fatigue. Scale score is the mean value of the nine items. When the total score is below 4, it is considered as "not tired" and when it is above 4, it is considered as "tired".
Rivermead Mobility Index | 12 week
  mobility.Total score is between 0-15. The score of 15 means that there is no problem in mobility, while a score of 14 and below means that there is a problem in mobility.
Functional Independence Scale | 12 week
  functional status.It consists of 18 items under six headings: self-care, sphincter control, transfer, displacement, communication and social perception. Every item is scored between 1-7 (1 point: fully dependent, 7 points: fully independent). It is possible to get a minimum score of 18 and a maximum score of 126.

CONTACTS AND LOCATIONS:
Overall Officials: Raziye Çelik, PT., Principal Investigator — Pamukkale University; Emre Baskan, Assoc Prof., Study Director — Pamukkale University; Aziz Dengiz, PT Phd, Study Director — Muş Alparslan University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known whether there will be a plan to roll out IPD.

REFERENCES:
- [Background] Sudlow CL, Warlow CP. Comparing stroke incidence worldwide: what makes studies comparable? Stroke. 1996 Mar;27(3):550-8. doi: 10.1161/01.str.27.3.550. PMID 8610328
- [Background] Kleindorfer DO, Towfighi A, Chaturvedi S, Cockroft KM, Gutierrez J, Lombardi-Hill D, Kamel H, Kernan WN, Kittner SJ, Leira EC, Lennon O, Meschia JF, Nguyen TN, Pollak PM, Santangeli P, Sharrief AZ, Smith SC Jr, Turan TN, Williams LS. 2021 Guideline for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021 Jul;52(7):e364-e467. doi: 10.1161/STR.0000000000000375. Epub 2021 May 24. No abstract available. PMID 34024117
- [Background] Siotto M, Germanotta M, Guerrini A, Pascali S, Cipollini V, Cortellini L, Ruco E, Khazrai YM, De Gara L, Aprile I. Relationship between Nutritional Status, Food Consumption and Sarcopenia in Post-Stroke Rehabilitation: Preliminary Data. Nutrients. 2022 Nov 15;14(22):4825. doi: 10.3390/nu14224825. PMID 36432512
- [Background] Purroy F, Montala N. Epidemiology of stroke in the last decade: a systematic review. Rev Neurol. 2021 Nov 1;73(9):321-336. doi: 10.33588/rn.7309.2021138. English, Spanish. PMID 34676530
- [Background] Scherbakov N, von Haehling S, Anker SD, Dirnagl U, Doehner W. Stroke induced Sarcopenia: muscle wasting and disability after stroke. Int J Cardiol. 2013 Dec 10;170(2):89-94. doi: 10.1016/j.ijcard.2013.10.031. Epub 2013 Oct 14. PMID 24231058
- [Background] Li S, Gonzalez-Buonomo J, Ghuman J, Huang X, Malik A, Yozbatiran N, Magat E, Francisco GE, Wu H, Frontera WR. Aging after stroke: how to define post-stroke sarcopenia and what are its risk factors? Eur J Phys Rehabil Med. 2022 Oct;58(5):683-692. doi: 10.23736/S1973-9087.22.07514-1. Epub 2022 Sep 5. PMID 36062331
- [Background] Su Y, Asamoto M, Yuki M, Saito M, Hasebe N, Hirayama K, Otsuki M, Iino C. Predictors and short-term outcomes of post-stroke fatigue in initial phase of transition from hospital to home: A prospective observational study. J Adv Nurs. 2021 Apr;77(4):1825-1838. doi: 10.1111/jan.14731. Epub 2020 Dec 23. PMID 33368578
- [Background] Paciaroni M, Acciarresi M. Poststroke Fatigue. Stroke. 2019 Jul;50(7):1927-1933. doi: 10.1161/STROKEAHA.119.023552. Epub 2019 Jun 14. No abstract available. PMID 31195940
- [Background] Mayo NE, Wood-Dauphinee S, Cote R, Durcan L, Carlton J. Activity, participation, and quality of life 6 months poststroke. Arch Phys Med Rehabil. 2002 Aug;83(8):1035-42. doi: 10.1053/apmr.2002.33984. PMID 12161823
- [Background] Tani Y, Otaka Y, Kudo M, Kurayama T, Kondo K. Prevalence of Genu Recurvatum during Walking and Associated Knee Pain in Chronic Hemiplegic Stroke Patients: A Preliminary Survey. J Stroke Cerebrovasc Dis. 2016 May;25(5):1153-1157. doi: 10.1016/j.jstrokecerebrovasdis.2016.01.028. Epub 2016 Feb 19. PMID 26907679
- [Background] Mally K, Trentmann J, Heller M, Dittmar M. Reliability and accuracy of segmental bioelectrical impedance analysis for assessing muscle and fat mass in older Europeans: a comparison with dual-energy X-ray absorptiometry. Eur J Appl Physiol. 2011 Aug;111(8):1879-87. doi: 10.1007/s00421-010-1795-x. Epub 2011 Jan 14. PMID 21234595
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Ozyemisci-Taskiran O, Batur EB, Yuksel S, Cengiz M, Karatas GK. Validity and reliability of fatigue severity scale in stroke. Top Stroke Rehabil. 2019 Mar;26(2):122-127. doi: 10.1080/10749357.2018.1550957. Epub 2018 Nov 26. PMID 30475156
- [Background] Collen FM, Wade DT, Robb GF, Bradshaw CM. The Rivermead Mobility Index: a further development of the Rivermead Motor Assessment. Int Disabil Stud. 1991 Apr-Jun;13(2):50-4. doi: 10.3109/03790799109166684. PMID 1836787
- [Background] Ottenbacher KJ, Hsu Y, Granger CV, Fiedler RC. The reliability of the functional independence measure: a quantitative review. Arch Phys Med Rehabil. 1996 Dec;77(12):1226-32. doi: 10.1016/s0003-9993(96)90184-7. PMID 8976303
- [Background] Chang KV, Wu WT, Huang KC, Han DS. Segmental body composition transitions in stroke patients: Trunks are different from extremities and strokes are as important as hemiparesis. Clin Nutr. 2020 Jun;39(6):1968-1973. doi: 10.1016/j.clnu.2019.08.024. Epub 2019 Aug 31. PMID 31522786
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Background] Ramsay JW, Barrance PJ, Buchanan TS, Higginson JS. Paretic muscle atrophy and non-contractile tissue content in individual muscles of the post-stroke lower extremity. J Biomech. 2011 Nov 10;44(16):2741-6. doi: 10.1016/j.jbiomech.2011.09.001. Epub 2011 Sep 25. PMID 21945568
- [Background] Borschmann K, Iuliano S, Ghasem-Zadeh A, Churilov L, Pang MYC, Bernhardt J. Upright activity and higher motor function may preserve bone mineral density within 6 months of stroke: a longitudinal study. Arch Osteoporos. 2018 Jan 8;13(1):5. doi: 10.1007/s11657-017-0414-4. PMID 29313169
- [Background] Aali G, Drummond A, das Nair R, Shokraneh F. Post-stroke fatigue: a scoping review. F1000Res. 2020 Apr 7;9:242. doi: 10.12688/f1000research.22880.2. eCollection 2020. PMID 32934800
- [Background] Choi-Kwon S, Choi SH, Suh M, Choi S, Cho KH, Nah HW, Song H, Kim JS. Musculoskeletal and central pain at 1 year post-stroke: associated factors and impact on quality of life. Acta Neurol Scand. 2017 Apr;135(4):419-425. doi: 10.1111/ane.12617. Epub 2016 Jun 6. PMID 27265610
- [Background] MacIntosh BJ, Edwards JD, Kang M, Cogo-Moreira H, Chen JL, Mochizuki G, Herrmann N, Swardfager W. Post-stroke Fatigue and Depressive Symptoms Are Differentially Related to Mobility and Cognitive Performance. Front Aging Neurosci. 2017 Oct 31;9:343. doi: 10.3389/fnagi.2017.00343. eCollection 2017. PMID 29163127
- [Background] Bye A, Sjoblom B, Wentzel-Larsen T, Gronberg BH, Baracos VE, Hjermstad MJ, Aass N, Bremnes RM, Flotten O, Jordhoy M. Muscle mass and association to quality of life in non-small cell lung cancer patients. J Cachexia Sarcopenia Muscle. 2017 Oct;8(5):759-767. doi: 10.1002/jcsm.12206. Epub 2017 May 10. PMID 28493418
- [Background] Wang B, Thapa S, Zhou T, Liu H, Li L, Peng G, Yu S. Cancer-related fatigue and biochemical parameters among cancer patients with different stages of sarcopenia. Support Care Cancer. 2020 Feb;28(2):581-588. doi: 10.1007/s00520-019-04717-0. Epub 2019 May 17. PMID 31102055
- [Background] al-Majid S, McCarthy DO. Cancer-induced fatigue and skeletal muscle wasting: the role of exercise. Biol Res Nurs. 2001 Jan;2(3):186-97. doi: 10.1177/109980040100200304. PMID 11547540
- [Background] Morgado PC, Giorlando A, Castro M, Navigante A. Relationship between weight loss and parameters of skeletal muscle function in patients with advanced cancer and fatigue. Support Care Cancer. 2016 Sep;24(9):3961-6. doi: 10.1007/s00520-016-3236-9. Epub 2016 Apr 28. PMID 27126771
- [Background] Neefjes ECW, van den Hurk RM, Blauwhoff-Buskermolen S, van der Vorst MJDL, Becker-Commissaris A, de van der Schueren MAE, Buffart LM, Verheul HMW. Muscle mass as a target to reduce fatigue in patients with advanced cancer. J Cachexia Sarcopenia Muscle. 2017 Aug;8(4):623-629. doi: 10.1002/jcsm.12199. Epub 2017 Jun 21. PMID 28639432
- [Background] Wagner LI, Cella D. Fatigue and cancer: causes, prevalence and treatment approaches. Br J Cancer. 2004 Aug 31;91(5):822-8. doi: 10.1038/sj.bjc.6602012. PMID 15238987
- [Background] Neefjes EC, van der Vorst MJ, Blauwhoff-Buskermolen S, Verheul HM. Aiming for a better understanding and management of cancer-related fatigue. Oncologist. 2013;18(10):1135-43. doi: 10.1634/theoncologist.2013-0076. Epub 2013 Sep 13. PMID 24037979
- [Background] Peters DM, O'Brien ES, Kamrud KE, Roberts SM, Rooney TA, Thibodeau KP, Balakrishnan S, Gell N, Mohapatra S. Utilization of wearable technology to assess gait and mobility post-stroke: a systematic review. J Neuroeng Rehabil. 2021 Apr 21;18(1):67. doi: 10.1186/s12984-021-00863-x. PMID 33882948
- [Background] Ursin MH, Ihle-Hansen H, Fure B, Tveit A, Bergland A. Effects of premorbid physical activity on stroke severity and post-stroke functioning. J Rehabil Med. 2015 Aug 18;47(7):612-7. doi: 10.2340/16501977-1972. PMID 26073856
- [Background] Hebert D, Lindsay MP, McIntyre A, Kirton A, Rumney PG, Bagg S, Bayley M, Dowlatshahi D, Dukelow S, Garnhum M, Glasser E, Halabi ML, Kang E, MacKay-Lyons M, Martino R, Rochette A, Rowe S, Salbach N, Semenko B, Stack B, Swinton L, Weber V, Mayer M, Verrilli S, DeVeber G, Andersen J, Barlow K, Cassidy C, Dilenge ME, Fehlings D, Hung R, Iruthayarajah J, Lenz L, Majnemer A, Purtzki J, Rafay M, Sonnenberg LK, Townley A, Janzen S, Foley N, Teasell R. Canadian stroke best practice recommendations: Stroke rehabilitation practice guidelines, update 2015. Int J Stroke. 2016 Jun;11(4):459-84. doi: 10.1177/1747493016643553. Epub 2016 Apr 14. PMID 27079654
- [Background] Silva CRRD, Pimenta CJL, Viana LRC, Ferreira GRS, Bezerra TA, Costa TFD, Pontes MLF, Costa KNFM. Specific health-related quality of life in Cerebrovascular accident survivors: associated factors. Rev Bras Enferm. 2021 Nov 29;75(3):e20210407. doi: 10.1590/0034-7167-2021-0407. eCollection 2021. English, Portuguese. PMID 34852127
- See also: Fitness ve EMS (Electromyostimulation) antrenman tekniklerinin vücut kompozisyonu üzerine etkileri — https://dergipark.org.tr/en/download/article-file/2232076
- See also: BF 1000 Super Pricision Kullanım Kılavuzu — https://www.kullanimkilavuzu.com.tr/beurer/bf-1000/k%C4%B1lavuz
- See also: Fazla kilolu ve obez kadınlarda 30 dakika egzersiz kilo kaybı üzerine etkili midir? — https://doi.org/10.30569/adiyamansaglik.739063
- See also: Rivermead mobilite indeksi (RMI) türkçe formunun yaşlılarda geçerlilik ve güvenilirliği — https://geriatri.dergisi.org/uploads/pdf/pdf_TJG_362.pdf
- See also: Türkiye'de nörorehabilitasyon hastalarının değerlendirilmesinde fonksiyonel bağımsızlık ölçeği ve Modifiye Barthel İndeksi'nin yeri — https://search.trdizin.gov.tr/tr/yayin/detay/12016/
- See also: Bone mineral density and its relationship with body composition indices in stroke patients — https://doi.org/10.22141/pjs.12.1.2022.322
- See also: İnme sonrası alt ekstremite, mobilite ve yürüme: alt ekstremite, hareketlilik ve inme sonrası yürüyüş. — https://dergipark.org.tr/tr/download/article-file/1088259
- See also: Impact of stroke on quality of life and functional independence:research article. — https://njppp.com/fulltext/28-1531996089.pdf